CLINICAL TRIAL: NCT02380001
Title: Analgesic Efficacy of Preoperative Oral Administration of Dexketoprofen Trometamol in Third Molar Surgery, Compared to Postoperative Administration
Brief Title: Analgesic Preoperative/Postoperative Dexketoprofen Trometamol in Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Chavarría Bolaños (Other)
Responsible Party: Sponsor-Investigator, Daniel Chavarría Bolaños, Dr. Daniel Chavarría Bolaños, MSc. PhD, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI-FE-028-014
Record Dates: First submitted 2015-02-22; First posted 2015-03-05 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Dexketoprofen trometamol; third molar surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexketoprofen trometamol (Experimental): A White round pill with 25 mg of dexketoprofen will be administered 30 minutes before the impacted third molar surgery start. Immediately after the surgery, a hard-gelatin capsule with placebo will be administered.
  Interventions: Drug: Dexketoprofen trometamol
- Preoperative control (Placebo Comparator): A hard-gelatin capsule with placebo will be administered 30 minutes before the impacted third molar surgery start. Immediately after the surgery, a hard-gelatin capsule with 25mg of Dexketoprofen will be administered.
  Interventions: Drug: Preoperative control

INTERVENTIONS:
Drug: Dexketoprofen trometamol — White round pill containing 25mg of Dexketoprofen will be administered either prior/after to third molar surgery.
  Other Names: Enantyum; Miracox
  Arms: Dexketoprofen trometamol
Drug: Preoperative control — white round pill containing 25mg of placebo will be administered prior/after to third molar surgery. The placebo pill is identical to active dexketoprofen, in size and color
  Other Names: Placebo
  Arms: Preoperative control

SUMMARY:
The purpose of the present investigation is to evaluate the effectiveness of the preoperative administration of Dexketoprofen Trometamol, employing the third molar surgery model, when compared to postoperative administration of the same drug. It was hypothesized that preoperative oral Dexketoprofen trometamol will reduce the intensity of pain by 30% after 8 hours of the surgery, when compared with post-operative administration.

DETAILED DESCRIPTION:
MODEL OF SURGICAL REMOVAL OF TOOTH IMPACTION. The model of Dental Impaction Pain Model (DIPM) is the most utilized of all the acute pain models. Its popularity is due to a well-established, well-validated, and extensively used postsurgery pain model in assessing the efficacy of analgesics on inflammatory pain.

The surgical procedure is very standardized and surgery require either minimal or nothing use of CNS depressant anesthetics. The methodology is similar to other models of acute pain; however, the DIPM is much more versatile than most other models. The model can be easily adapted to carry out studies of multiple-dose, pharmacokinetics / pharmacodynamics, preventive interventions and analgesic efficacy

The impacted lower third molar extraction involves the manipulation of hard and soft tissue, making the patient undergoes a series of effects which include acute pain, inflammation and trismus in the immediate postoperative period and goes from 24 to 72 postoperative hours. The pain associated with the surgical removal of a third molar is moderate to severe, increasing with greater intensity during the first 24 hours after surgery with spikes of pain between the first six to eight hours when using a conventional local anesthetic.

In this context, the control of pain and inflammation post-surgical associated with third molar removal has been very varied; highlighting the use of anti-inflammatory pain relievers non (NSAIDs) and some opioids.

PAIN. Pain is defined as the perception of a potentially injurious stimulus; which jointly to several not pleasurable experiences (sensory, emotional and cognitive), same that are caused by tissue damage (actual, potential or described in terms of such damage) and manifested by certain reactions physiological, autonomic and behavioral. Pain is typically classified as either acute or chronic.

Acute pain: is of sudden onset and is usually the result of a clearly defined cause such as an injury. The acute pain includes the estimated time as necessary so that the tissues heal, as described by John Bonica in 1953, usually in the span of a month, according to the Committee of taxonomy of the pains of IASP, the length limit for a sharp pain is three months, however should be noted that there are authors who continue classifying pain acute with a duration of up to 6 months.

Chronic pain: is defined as pain that lasts more than 12 weeks, or the one that according to the characteristics of their origin, exceeds time which could usually be defined a similar pain. It is accompanied by psychological commitment to important behavior disorders that can lead to depressive states; depending on the individual baseline emotional.

Although it can also be classified according to their structure (somatic or visceral) origin and physiological mechanism (nociceptive or neuropathic).

The scheme to perceive pain needs: a) a peripheral structure that acts as a receiver; b) a synapse in the spinal cord, c) pathways from spinal cord to superiority centers and d) descending pathways from the superiority center to the marrow, which act as mainly inhibitory mechanisms but also facilitated by change of neurotransmitters .

The study of the neurophysiology of pain has been an important advance in the knowledge of the mechanism of the painful stimulus in the perioperative period describing a dynamic system where multiple input have a place nociceptive, which conditions the first stage of peripheral awareness that amplifies transmission of stimulation to condition a second tier of central sensitization to keep in time.

MEASUREMENT OF PAIN. Clinicians and researchers have recognized that pain is a multidimensional experience, which includes a number of qualities or measurable elements as intensity, involvement, sensory quality, quality spatial (location), temporary quality, and the impact on daily activities. While the focus on the measurement of pain remain in the intensity, there has been an increase in the interest of measure other elements of pain.

PAIN INTENSITY SCALES. The domain of pain used in clinical studies and research is the intensity of the pain. The three scales used to measure the intensity of pain are: a) visual analog (VAS scale), b) the scale of numeric value (NRS) and c) the verbal value (VRS).

STRATEGIES IN THE MANAGEMENT OF DENTAL PAIN.

In dental practice pain of moderate to severe intensity conditions are usually treated with Nonstereoidal anti-inflammatory (NSAIDs) drug, although there are other different types of drugs used for this purpose that are described below:

* NASAIDs are a class of drugs that provides analgesic and antipyretic effects. Since they have a mechanism of action in common based on the inhibition of cyclooxygenase (COX) enzyme responsible for the biosynthesis of prostaglandins and general of Eicosanoids. Unfortunately, prostaglandins mediate other physiological functions that cause undesirables adverse effects.
* New inhibitors of COX show great power and analgesic effectiveness and are better at reducing the incidence of adverse effects compared to the classic AINE´S.

DEXKETOPROFEN TROMETAMOL. Dexketoprofen is a new anti-inflammatory drug non-steroidal (NSAID) belonging to the family of the arylpropionic acid derivatives. Dexketoprofen is the enantiomer S (+) of the composite ketoprofen, a drug with analgesic effects and anti-inflammatory clearly documented.

Dexketoprofen has been developed (dexketoprofen trometamol) tromethamine salt as a formulation with a higher than the free acid aqueous solubility. Pharmacokinetic studies performed in healthy individuals showed that oral administration of dexketoprofen trometamol presented a kinetic favorable profile for use in acute pain compared to the formulation of free acid or racemic ketoprofen.

Dexketoprofen trometamol, is one of the most powerful inhibitors of prostaglandin synthesis "in vitro". 12.5-25 mg orally is given with a quickly absorbed on an empty stomach, which has a strong binding to albumin and inactive metabolites after glucuronization renal excretion. It is well accumulate in synovial fluid and its analgesic potency is comparable to 50 mg of ketoprofen or diclofenac and more than 600 mg of ibuprofen, so its main indication is acute postoperative pain.

The production of a unique isomer of ketoprofen formulation simplifies the pharmacokinetics of the drug and allows a reduction of 50% in the dose. This can reduce adverse effects to reduce the metabolic and renal work, rapid absorption appears to offer some protection against gastrointestinal complications as a method to avoid gastrointestinal toxicity different of the selectivity of COX presents a good profile of security and reported adverse effects are similar to placebo in these studies, the uniqueness of the therapeutic profile of the DKP.TRIS could be the result of a combination of factors which include the higher power as it is given only the active molecule, inhibition of COX two isoenzymes, rapid absorption from the gastrointestinal tract and high capacity to enter the CNS.

PREVENTIVE ANALGESIA. Preventive analgesia (PA) is an antinociceptive treatment which prevents the establishment of the altered processing of the sensory input, that amplifies and chronic postoperative pain. The PA concept was formulated by Crile at the beginning of the century on the basis of clinical observations. There are two terms in English which refer to the same concept: preemptive analgesia, which consists of a treatment that is given before the surgical incision and maintained for intervention to avoid an altered sensory processing that amplifies and chronic postoperative pain. Is usually to compare the same way and the same drug management before and after the incision; and preventive analgesia consists of a longer lasting analgesic effect which that would theoretically be expected after administration of a certain drug on the basis of its pharmacological properties.

In oral surgery, primary hyperalgesia is the awareness of the receivers of the mucosa and the periosteum by a range of mediators of inflammation such as prostaglandins. Secondary hyperalgesia is central sensitization of neurons in the nucleus trigeminal and spinal supra structures. Secondary hyperalgesia can be observed over the time, while the primary hyperalgesia is provable within a few hours after the injury; Prostaglandins are synthesized quickly after damage to the tissue and appear in significant concentrations 1 hour after trauma.

The concept of preventive analgesia is based on the prior administration to the surgical incision of a painkiller to dampen or prevent phenomena of hypersensitisation central in order to reduce the consumption of analgesics in the postoperative period.

WORK PLAN. Using a format in which specify the inclusion and exclusion criteria, the selection of the patients will be held, during this visit will also fill the form of demographic data, status of the patient, current condition, medical history, physical examination, x-ray and diagnostic studies. See annex 3.

Then patients will be randomized distributed in two groups of participants, group 1 and 2:

Experimental drugs. The randomized patient is determined to a group according with the administration of the drug in two groups.

GROUP 1 Oral administration of dexketoprofen Trometamol 25 mg, 30 minutes before the beginning of surgery and administered immediately at the end of the same placebo.

GROUP 2 The placebo is oral administered 30 minutes before the beginning of surgery and administered immediately at the end of the same dexketoprofen Trometamol 25 mg.

Surgical procedure. All surgeries will be performed by the same surgeon, to achieve a local anesthetic effect, a previous asepsis and antisepsis of the area will be necessary. The lower alveolar nerve with reinforcement of the lingual nerve and long buccal nerve using 2 cartridges of lidocaine with epinephrine 2% with a concentration of 1:100 ml.

Once the anaesthetic effect is present, surgery can be performed, a flap of total thickness of mucoperiosteal will be made, using a triangular incision design liberating the tissue at the level of the second mandibular molar, subsequently the third molar extraction will be performed. Finally the reposition of the flap and suturing will be made using black silk suture (3-0).

In all cases the duration of the surgery procedure will be registered in every step. see annex 4.

Measurement of the variables. Intensity of pain. For both groups, a measure will be performed between the distance in mm from point 0 to the point that the patient indicates; with the understanding that the point represents the intensity of the pain using the NRS, values were registered in the NRS scale of each patient. This procedure will beginning after the second intake of the drug or placebo (basal), after 8 hours (8-NRS), 24 hours, 48 hours and 72 hours post operatory.

Time to remedication. The time in minutes that the patient request remedication with dexketoprofen, registering again the intensity of pain will be registered.

Total of tablets consumed. The number of tablets consumed in the 72 hrs of the postoperative will be recorded. The dosage of dexketoprofen 25mg will be standardized for every 8 hours, and not to exceed 75mg every 24 hours until the patient deems necessary.

The antibiotic used in the clinical trial will be:

Clindamycin 300 mg every 8 hrs for 5 days. After 7 days of postoperative evolution, the patient will return to the clinic for removal of stitches, evaluating the operative area and general health condition, with this step, the attention will be concluded for the surgical procedure and the medical discharge will be indicated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18-28 years old
* Clinical and radiographic diagnosis of impacted mandibular third molars, which the surgical approach may include flap and osteotomy procedures.
* surgery classified as simple to moderate
* Voluntary acceptance of written consent, previously approved by institutional ethics committee

Exclusion Criteria:

* Prior administration of analgesic or anti-inflammatory drugs
* History of drug dependence
* History of allergic reactions to any of the drugs selected, or local anesthetics
* Simultaneous presence of oral pathologies that may interfere with the surgical procedure

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain measurement employing a previous validated visual analogue scale of pain (VAS). | 72 hours
  Postoperative pain measurement will be held every 8 hours for the next 72 hours after the surgical intervention

SECONDARY OUTCOMES:
Number of patients with adverse events, to determine tolerability of the drugs. | 7 days
  immediate after the surgery is completed, and for the next 7 days, any adverse reaction will be recorded
needing of second dosage administration | 72 hours
  After the immediate administration of Dexketoprofen once the surgery is completed, the number of new doses needed will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amaury Pozos, PhD, Study Director — Universidad Autonoma de San Luis Potosí; Vicente Esparza, Resident, Principal Investigator — Universidad Autonoma de San Luis Potosí
Locations (1):
- FACULTY OF MEDICINE, San Luis Potosi University, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Cooper SA, Desjardins PJ. The value of the dental impaction pain model in drug development. Methods Mol Biol. 2010;617:175-90. doi: 10.1007/978-1-60327-323-7_15. PMID 20336423
- [Background] Marciani RD. Third molar removal: an overview of indications, imaging, evaluation, and assessment of risk. Oral Maxillofac Surg Clin North Am. 2007 Feb;19(1):1-13, v. doi: 10.1016/j.coms.2006.11.007. PMID 18088860
- [Background] Seymour RA, Meechan JG, Blair GS. An investigation into post-operative pain after third molar surgery under local analgesia. Br J Oral Maxillofac Surg. 1985 Dec;23(6):410-8. doi: 10.1016/0266-4356(85)90025-7. PMID 2933061
- [Background] Pozos AJ, Martinez R, Aguirre P, Perez J. Tramadol administered in a combination of routes for reducing pain after removal of an impacted mandibular third molar. J Oral Maxillofac Surg. 2007 Aug;65(8):1633-9. doi: 10.1016/j.joms.2006.06.267. No abstract available. PMID 17656294
- [Background] Isiordia-Espinoza MA, Pozos-Guillen AJ, Martinez-Rider R, Herrera-Abarca JE, Perez-Urizar J. Preemptive analgesic effectiveness of oral ketorolac plus local tramadol after impacted mandibular third molar surgery. Med Oral Patol Oral Cir Bucal. 2011 Sep 1;16(6):e776-80. doi: 10.4317/medoral.16854. PMID 21217614
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Barden J, Edwards JE, McQuay HJ, Wiffen PJ, Moore RA. Relative efficacy of oral analgesics after third molar extraction. Br Dent J. 2004 Oct 9;197(7):407-11; discussion 397. doi: 10.1038/sj.bdj.4811721. PMID 15475903
- [Background] Gajraj NM, Joshi GP. Role of cyclooxygenase-2 inhibitors in postoperative pain management. Anesthesiol Clin North Am. 2005 Mar;23(1):49-72. doi: 10.1016/j.atc.2004.11.011. PMID 15763411
- [Background] Coxib and traditional NSAID Trialists' (CNT) Collaboration; Bhala N, Emberson J, Merhi A, Abramson S, Arber N, Baron JA, Bombardier C, Cannon C, Farkouh ME, FitzGerald GA, Goss P, Halls H, Hawk E, Hawkey C, Hennekens C, Hochberg M, Holland LE, Kearney PM, Laine L, Lanas A, Lance P, Laupacis A, Oates J, Patrono C, Schnitzer TJ, Solomon S, Tugwell P, Wilson K, Wittes J, Baigent C. Vascular and upper gastrointestinal effects of non-steroidal anti-inflammatory drugs: meta-analyses of individual participant data from randomised trials. Lancet. 2013 Aug 31;382(9894):769-79. doi: 10.1016/S0140-6736(13)60900-9. Epub 2013 May 30. PMID 23726390
- [Background] Hawkey CJ. COX-1 and COX-2 inhibitors. Best Pract Res Clin Gastroenterol. 2001 Oct;15(5):801-20. doi: 10.1053/bega.2001.0236. PMID 11566042
- [Background] Jin F, Chung F. Multimodal analgesia for postoperative pain control. J Clin Anesth. 2001 Nov;13(7):524-39. doi: 10.1016/s0952-8180(01)00320-8. PMID 11704453
- [Background] Rodriguez MJ, Arbos RM, Amaro SR. Dexketoprofen trometamol: clinical evidence supporting its role as a painkiller. Expert Rev Neurother. 2008 Nov;8(11):1625-40. doi: 10.1586/14737175.8.11.1625. PMID 18986233
- [Background] Veys EM. 20 years' experience with ketoprofen. Scand J Rheumatol Suppl. 1991;90:Suppl 1-44. PMID 1947892
- [Background] Mauleon D, Artigas R, Garcia ML, Carganico G. Preclinical and clinical development of dexketoprofen. Drugs. 1996;52 Suppl 5:24-45; discussion 45-6. doi: 10.2165/00003495-199600525-00005. PMID 8922555
- [Background] Barbanoj MJ, Antonijoan RM, Gich I. Clinical pharmacokinetics of dexketoprofen. Clin Pharmacokinet. 2001;40(4):245-62. doi: 10.2165/00003088-200140040-00002. PMID 11368291
- [Background] Katz J, Clarke H, Seltzer Z. Review article: Preventive analgesia: quo vadimus? Anesth Analg. 2011 Nov;113(5):1242-53. doi: 10.1213/ANE.0b013e31822c9a59. Epub 2011 Sep 30. PMID 21965352
- [Background] Savage MG, Henry MA. Preoperative nonsteroidal anti-inflammatory agents: review of the literature. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Aug;98(2):146-52. doi: 10.1016/j.tripleo.2004.01.012. PMID 15316540
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Kelly DJ, Ahmad M, Brull SJ. Preemptive analgesia I: physiological pathways and pharmacological modalities. Can J Anaesth. 2001 Nov;48(10):1000-10. doi: 10.1007/BF03016591. PMID 11698320
- [Background] Moiniche S, Kehlet H, Dahl JB. A qualitative and quantitative systematic review of preemptive analgesia for postoperative pain relief: the role of timing of analgesia. Anesthesiology. 2002 Mar;96(3):725-41. doi: 10.1097/00000542-200203000-00032. No abstract available. PMID 11873051
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Kissin I. Preemptive analgesia. Anesthesiology. 2000 Oct;93(4):1138-43. doi: 10.1097/00000542-200010000-00040. No abstract available. PMID 11020772
- [Background] Dahl JB, Moiniche S. Pre-emptive analgesia. Br Med Bull. 2004 Dec 13;71:13-27. doi: 10.1093/bmb/ldh030. Print 2004. PMID 15596866
- [Background] Brennan TJ, Kehlet H. Preventive analgesia to reduce wound hyperalgesia and persistent postsurgical pain: not an easy path. Anesthesiology. 2005 Oct;103(4):681-3. doi: 10.1097/00000542-200510000-00004. No abstract available. PMID 16192759
- [Background] Kissin I. Preemptive analgesia at the crossroad. Anesth Analg. 2005 Mar;100(3):754-756. doi: 10.1213/01.ANE.0000144429.39988.9B. No abstract available. PMID 15728065
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Vadivelu N, Mitra S, Schermer E, Kodumudi V, Kaye AD, Urman RD. Preventive analgesia for postoperative pain control: a broader concept. Local Reg Anesth. 2014 May 29;7:17-22. doi: 10.2147/LRA.S62160. eCollection 2014. PMID 24872720
- [Background] Sagiroglu G. Comparing early postoperative period analgesic effect of dexketoprofene trometamol and lornoxicam in mediastinoscopy cases. Eurasian J Med. 2011 Apr;43(1):23-6. doi: 10.5152/eajm.2011.05. PMID 25610155
- [Background] Kara I, Tuncer S, Erol A, Reisli R. [The effects of preemptive dexketoprofen use on postoperative pain relief and tramadol consumption]. Agri. 2011 Jan;23(1):18-21. doi: 10.5505/agri.2011.21939. Turkish. PMID 21341148
- [Background] Kesimci E, Gumus T, Izdes S, Sen P, Kanbak O. Comparison of efficacy of dexketoprofen versus paracetamol on postoperative pain and morphine consumption in laminectomy patients. Agri. 2011 Oct;23(4):153-9. doi: 10.5505/agri.2011.86548. PMID 22290679
- [Background] Cagiran E, Eyigor C, Sezer B, Uyar M. Preemptive analgesic efficacy of dexketoprofen trometamol on impacted third molar surgery. Agri. 2014;26(1):29-33. doi: 10.5505/agri.2014.55265. PMID 24481581
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Juodzbalys G, Daugela P. Mandibular third molar impaction: review of literature and a proposal of a classification. J Oral Maxillofac Res. 2013 Jul 1;4(2):e1. doi: 10.5037/jomr.2013.4201. PMID 24422029
- [Derived] Esparza-Villalpando V, Chavarria-Bolanos D, Gordillo-Moscoso A, Masuoka-Ito D, Martinez-Rider R, Isiordia-Espinoza M, Pozos-Guillen A. Comparison of the analgesic efficacy of preoperative/postoperative oral dexketoprofen trometamol in third molar surgery: A randomized clinical trial. J Craniomaxillofac Surg. 2016 Sep;44(9):1350-5. doi: 10.1016/j.jcms.2016.06.002. Epub 2016 Jun 9. PMID 27378000